CLINICAL TRIAL: NCT06794866
Title: A Phase 3, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Safety and Efficacy of OnabotulinumtoxinA Purified Neurotoxin Complex for the Treatment of Moderate to Severe Forehead Lines in Japan
Brief Title: A Study to Assess Adverse Events and Effectiveness of OnabotulinumtoxinA Intramuscular Injections for the Change of Moderate to Severe Forehead Lines in Adult Participants
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M24-697
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Forehead Lines
Keywords: Forehead Lines; OnabotulinumtoxinA; FHL Japan P3
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1 (Experimental): Participants will receive onabotulinumtoxinA Dose A in both Period 1 and Period 2.
  Interventions: Drug: OnabotulinumtoxinA
- Group 2 (Experimental): Participants will receive onabotulinumtoxinA Dose B in both Period 1 and Period 2.
  Interventions: Drug: OnabotulinumtoxinA
- Group 3 (Experimental): Participants will receive placebo in Period 1 and onabotulinumtoxinA Dose A in Period 2.
  Interventions: Drug: OnabotulinumtoxinA; Drug: Placebo
- Group 4 (Experimental): Participants will receive placebo in Period 1 and onabotulinumtoxinA Dose B in Period 2.
  Interventions: Drug: OnabotulinumtoxinA; Drug: Placebo

INTERVENTIONS:
Drug: OnabotulinumtoxinA — Intramuscular Injections
Drug: Placebo — Intramuscular Injections
  Arms: Group 3; Group 4

SUMMARY:
Facial lines that develop from repeated facial expression, such as forehead lines (FHL), are typically treated by selectively weakening specific muscles with small quantities of botulinum toxin. The purpose of this study is to assess adverse events and effectiveness of onabotulinumtoxinA in Japanese adults with moderate to severe FHL.

Participants are placed in 1 of 4 groups, called treatment arms. Each group receives a different treatment. Participants are randomly assigned to receive onabotulinumtoxinA or placebo. There is a 1 in 5 chance that a participant will receive placebo. Around 150 adult participants with moderate to severe FHL will be enrolled in the study in approximately 15 sites in Japan.

In Period 1, participants will receive intramuscular injections on Day 1. In Period 2, participants will receive up to 3 additional treatment cycles. Participants will be followed for up to 12 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at the study site. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Forehead lines (FHL) of moderate or severe rating at maximum contraction as assessed by investigator using the Facial Wrinkle Scale with Asian Photonumeric Guide (FWS-A) at Day 1 prior to study treatment.
* Glabellar lines (GL) of moderate or severe rating at maximum contraction as assessed by investigator using the FWS-A at Day 1 prior to study treatment.
* Good health as per the investigator's judgment based on medical history, abbreviated physical examination and vital sign measurements, including no known active pandemic infection (e.g., severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2]).

Exclusion Criteria:

* FHL of severe rating at rest as assessed by investigator using the FWS-A at Day 1 prior to study treatment.
* History of known immunization or hypersensitivity to any botulinum neurotoxin serotype.
* History of treatments to the mid or upper face.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve 'None' or 'Mild' on Facial Wrinkle Scale with Asian Photonumeric Guide (FWS-A) According to the Investigator Assessment of Forehead Lines (FHL) Severity at Maximum Contraction | Day 30
  The investigator assesses FHL severity using the FWS-A scale ranging from none to severe.
Number of Participants with Adverse Events (AEs) | Up to approximately 12 months
  Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants who Achieved 'None' or 'Mild' on FWS-A According to the Participant Assessment of FHL Severity | Day 30
  The participant assesses FHL severity using the FWS-A scale ranging from none to severe.
Percentage of Participants who Achieved at least 1-Grade Improvement from Baseline on FWS-A According to the Investigator Assessment of FHL Severity at Maximum Contraction | Day 30
  The investigator assesses FHL severity using the FWS-A scale ranging from none to severe.
Percentage of Participants who Achieved at least 1-Grade Improvement from Baseline on FWS-A According to the Investigator Assessment of FHL Severity at Rest | Day 30
  For participants rated as at least mild at baseline, the investigator assesses FHL severity using the FWS-A scale ranging from none to severe.
Time to Return to at least 'Moderate' for the Participants who Achieve Investigator FWS-A ratings of 'None' or 'Mild' on FHL Severity at Maximum Contraction | Day 30
  The investigator assesses FHL severity using the FWS-A scale ranging from none to severe.
Percentage of Participants with Responder Status of 'Very Satisfied' or 'Mostly Satisfied' on Satisfaction with Treatment on the Facial Line Satisfaction Questionnaire (FLSQ) | Day 60
  The FLSQ assesses treatment satisfaction and psychosocial impact. Participants assessed their satisfaction with FHL using the FLSQ scale ranging from Very dissatisfied to Very satisfied.
Percentage of Participants with Responder Status of 'Very Satisfied' or 'Mostly Satisfied' on Satisfaction with Natural Look on the FLSQ | Day 30
  The FLSQ assesses treatment satisfaction and psychosocial impact. Participants assessed their satisfaction with FHL using the FLSQ scale ranging from Very dissatisfied to Very satisfied.
Change from Baseline in the Participant's Rasch-Transformed Score of the SKIN-Q Scale | Day 30
  The SKIN-Q Scale is a scale that measures the appearance of skin quality response option ranging from Very dissatisfied to Very satisfied.
Change from Baseline in the Participant's Rasch-Transformed Score of the FACE-Q Social Function Scale at the Final Visit | Day 30
  The FACE-Q Psychological Function is a scale that measures psychological function with options ranging from definitely disagree to definitely agree.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (15):
- Japan (15):
  - Hiroshima Station Clinic /ID# 268467, Hiroshima, Hiroshima
  - Kotoni Tower Skin And Cosmetic Surgery Clinic /ID# 268460, Sapporo, Hokkaido
  - Tokai University Hospital /ID# 268496, Isehara, Kanagawa
  - Queen's Square Medical Center, Dermatology and Allergology /ID# 268454, Yokohama, Kanagawa
  - Jun Clinic /ID# 268531, Nagano, Nagano
  - Touyama Plastic Surgery Clinic /ID# 268456, Naha, Okinawa
  - Yoshikawa Skin Clinic /ID# 268494, Takatsuki, Osaka
  - Tokyo Center Clinic /ID# 268477, Chuo-ku, Tokyo
  - Tokyo Asbo Clinic /ID# 268529, Chuo-ku, Tokyo
  - Ginza Skin Clinic /ID# 268532, Chuo-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 268499, Minato-ku, Tokyo
  - Forest Palace Dermatology Clinic /ID# 268599, Nerima-ku, Tokyo
  - Greenwood skin clinic Tachikawa /ID# 268528, Tachikawa-shi, Tokyo
  - Chiharu Dermatology Clinic Urawa /ID# 268497, Saitama
  - Akihabara Skin Clinic /ID# 268441, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-697